CLINICAL TRIAL: NCT05548361
Title: The Use of Chlorhexidine and a Probiotic Lozenge in the Nonsurgical Therapy of Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Collaborators: BioGaia AB (Industry); Sunstar (Unknown)
Responsible Party: Principal Investigator, Mustafa Ozcan, Associate professor, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CukurovaU-PerII
Record Dates: First submitted 2022-09-12; First posted 2022-09-21 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Periodontitis; Chlorhexidine; Probiotic
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Active Chx (Experimental): This group will receive active chlorhexidine and placebo probiotics
  Interventions: Combination Product: active chlorhexidine and placebo probiotic
- Active probiotics (Experimental): This group will receive placeo chlorhexidine and active probiotics
  Interventions: Combination Product: placebo chlorhexidine and active probiotic
- Active Chx & probiotics (Experimental): This group will receive active chlorhexidine and active probiotics
  Interventions: Combination Product: active chlorhexidine and active probiotic

INTERVENTIONS:
Combination Product: active chlorhexidine and placebo probiotic — the randomized patients will be receive active chlorhexidine rinse and placebo probiotic
  Arms: Active Chx
Combination Product: placebo chlorhexidine and active probiotic — the randomized patients will receive placebo chlorhexidine rinse and active probiotic
  Arms: Active probiotics
Combination Product: active chlorhexidine and active probiotic — the randomized patients will receive active chlorhexidine rinse and active probiotic
  Arms: Active Chx & probiotics

SUMMARY:
The aim of this study is determining the additional effect of a 2-week home usage of chlorhexidine in periodontitis patients undergoing scaling and root planing supplemented with a dual-strain probiotic lozenge.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with generalized (>30% of teeth affected) periodontitisstage III and IV periodontitis, grade B or C (C only with smoker modifier) = generalized chronic periodontitis including smokers
* A minimum of three natural teeth in each quadrant, excluding third molars
* Willing and able to give informed consent
* Not more than 50% of the patients in each group will be smokers.
* Smokers should smoke between 10 to 40 cigarettes a day

Exclusion Criteria:

* Patients with localized periodontitis or periodontitis stage I or II or grade A or grade C or grade C with diabetes modifier
* Patients with orthodontic appliances (removable or fixed)
* Pregnant or lactating woman
* Patients with a history of systemic diseases that may correlate with periodontal health, such as diabetesrheumatic fever, liver or kidney disease, and neurological deficiencies
* Patients taking medication which may affect the periodontium (bisphosphonates, phenytoin, cyclosporin, nifidepine, chronic use of non-steroidal anti-inflammatory drugs)
* Patient who had taken systemic antibiotics up to 3 months prior to treatment or medical conditions requiring prophylactic antibiotic coverage
* Participation in any other clinical study
* Tobacco chewing or sniffing

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
probing pocket depth | 6 months
  the distance between gingival margin and pocket base in millimeters

SECONDARY OUTCOMES:
percentage of patients in low risk for disease progression | 6 months
  having less than 5 sites with probing pocket depth of 5 mm or more at the end of the trial.
gingival recession | 6 months
  the distance between cementoenamel junction and gingival margin in millimeters
clinical attachment level | 6 months
  the distance between cementoenamel junction and pocket base in millimeters
full mouth bleeding and plaque score | 6 months
  the scores of bleeding on probing (positive or negative)
microbial outcomes | 6 months
  pcr analysis of plaque samples (mean log10 cfg/ml)

CONTACTS AND LOCATIONS:
Locations (1):
- Cukurova university Faculty of Dentistry, Adana, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided